CLINICAL TRIAL: NCT00429715
Title: A Randomized, Safety, Immunogenicity & Efficacy Study of Autoclaved Leishmania Major Plus BCG vs. BCG (Double Blind) or Placebo (Open), in Healthy High Risk Iranian Volunteers With no Response to Leishmanin
Brief Title: Safety/Efficacy Trial of Killed Leishmania Vaccine in Volunteers With no Response to Leishmanin
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: Pasteur Institute of Iran, Tehran, Iran (Unknown); Razi Vaccine and Serum Research Institute (Other); Centre for Disease Control & Management, Ministry of Health & Medical Education (Other Government)
Responsible Party: Ali Khamesipour, Associate Professor, Center for Research & Training in Skin Diseases & Leprosy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CT110-1384; J/423/1057, 30/05/1385
Record Dates: First submitted 2007-01-31; First posted 2007-02-01 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2011-02

CONDITIONS: Healthy
Keywords: Leishmaniasis vaccine; Alum-ALM; First generation vaccine; Healthy volunteers; No response to leishmanin; No history of cutaneous leishmaniasis

ARMS (3):
- Alum-ALM + BCG (Experimental): Alum-ALM + BCG
  Interventions: Biological: Alum-ALM + BCG
- BCG (Active Comparator): BCG
  Interventions: Biological: Alum-ALM + BCG
- BCG diluent (Placebo Comparator): Diluent
  Interventions: Biological: Alum-ALM + BCG

INTERVENTIONS:
Biological: Alum-ALM + BCG — Alum precipitated autoclaved L. major
  Other Names: Alum precipitated autoclaved L. major
Biological: Alum-ALM + BCG — Arm 1=Alum-ALM + BCG Arm 2=BCG Arm 3=Placebo comparator
Biological: Alum-ALM + BCG — Alum-ALM + BCG

SUMMARY:
Development of a safe and effective vaccine against leishmaniasis started more than 10 years ago under WHO/TDR supervision. An autoclaved L. major vaccine (ALM) mixed with BCG has been tested in human in Iran, Pakistan and Sudan. Long term follow up of the vaccinees showed no untoward reactions except the skin reaction at the site of injection. The efficacy results of ALM was not satisfactory. In order to enhance immunogenicity of the vaccine, ALM was adsorbed to alum (Aluminum hydroxide). Alum-ALM plus adjuvant showed to induce protection in Rhesus monkeys against cutaneous leishmaniasis and in Languor monkeys against visceral leishmaniasis. Two trials of a single injection of different doses of Alum-ALM mixed with 1/10th of normal dose of BCG was carried out in healthy volunteers from a non endemic area of Sudan. The safety/immunogenicity parameters of the volunteers were closely monitored and the results showed that side effects were minimal and confined to the site of injection in the form of mild local pain, induration and ulceration, all associated with BCG vaccination. The immunogenicity results showed the strongest immune response seen in any Leishmania vaccine trials so far. It seems that this new formulation is an appropriate candidate for further development. Inoculation with live virulent Leishmania to produce a lesion for the purpose of preventing natural infection is known as leishmanization. The induced lesion heals and the person is usually protected against further infections. This method of prevention was practiced for centuries in the region. In this study volunteers with no response to leishmanin will be injected twice (30 days apart) with Alum-ALM 200 ug + 1/10 of BCG (n = 50) or BCG (n = 50) or BCG diluent alone (n = 50) as control. All volunteers will be leishmanized on day 60 post vaccination. In this trial, volunteers are protected either by vaccine or by leishmanization. The leishmanized volunteers will be visited by weekly and the development and healing process of the lesion will be monitored until complete healing of every volunteer. The immune responses of the volunteers will be evaluated. Vaccine efficacy is defined by the percent reduction in the number of volunteers developing a lesion following leishmanization as compared to controls on days 240.

DETAILED DESCRIPTION:
Background Information Leishmaniases encompass diverse clinical manifestations produced by different species of the protozoan parasite, Leishmania, transmitted by the bites of infected female sand flies. Due to the diversity of epidemiological characteristics, vector and reservoir control are impractical, costly and usually require political environment and infrastructures beyond the means of the countries suffering most from this disease. It was the aim of WHO/TDR to develop a safe and effective vaccine, which can be locally produced and thereby affordable for the populations of the poorest developing countries.

Beginning in the 1930's and 40's, Latin American scientists used killed whole parasite as a vaccine against leishmaniasis (1). Different forms of the vaccine, with or without adjuvant for prophylaxis or therapy have been studied in several countries in the past few decades (2), none has been efficacious for prophylaxis, but efficacy has been observed for immuno-chemotherapy (3). Over the past decade, we have produced and tested different preparations of killed L. major plus BCG. The autoclaved L. major (ALM) mixed with BCG (1/10th of the dose normally used as a vaccine against tuberculosis) was studied extensively in several clinical trials. The ALM + BCG formulation was shown to be safe and immunogenic (4-8). However, results from several phase III trials with a single or double-dose of this candidate vaccine against CL or VL did not show significant overall protection compared to immunization with BCG alone (6-8). Even three injections were not sufficiently protective against cutaneous leishmaniasis (CL).

In order to enhance immunogenicity of ALM + BCG, ALM was adsorbed to alum (Aluminum hydroxide), and the resulting alum-ALM was mixed with BCG to produce a new formulation for this vaccine. Indeed, the addition of alum to ALM leads to enhanced immunogenicity. It was demonstrated that a single injection of ALM in alum plus IL-12 induced protection in Rhesus monkeys against CL (10). Likewise, Alum-ALM + BCG protected Langur monkeys against visceral leishmaniasis (11).

The results of 2 dose escalating trials of a single intra-dermal injection of Alum-ALM (10 - 400 ug of Leishmania proteins) mixed with 1/10th normal dose of BCG showed the highest skin test conversion seen in any Leishmania vaccine trials so far (12). The safety parameters of the volunteers were closely monitored for 90 days after vaccination for local and systemic side effects. Side effects were minimal and confined to the site of injection. No systemic side effect was recorded. In the second TDR-sponsored trial in Sudan 10, 100 and 320 ug of the protein plus BCG were tested with results confirming the immunogenicity of the alum-ALM+BCG vaccine. Thus, Alum precipitated ALM mixed with 1/10th of BCG appears to constitute a safe vaccine and an appropriate candidate for further development.

Leishmanization (LZ):

Inoculation with live virulent Leishmania to produce a lesion for the purpose of preventing natural infection - which usually results in multiple lesions on exposed parts of the body - is known as leishmanization (LZ). Generally, recovery from CL leads to protection against future infection (14). During the last forty years, L. major promastigotes grown in cell-free culture have been used for leishmanization in Israel (15) and Iran (16) as well as in a high-risk population in Uzbekistan (17). Massive LZ was performed on an estimated two million people in Iran as a preventive measure during the Iran-Iraq war in the 80's (16). However, this practice was discontinued after the war due to occasional long-lasting lesions and the difficulties of standardized production under the circumstances immediately following the war.

LZ as a live challenge in efficacy trials of leishmaniasis candidate vaccines would bring about considerable time and cost saving by dramatically reducing the follow-up time, logistical demands and sample size required (thereby exposing fewer participants to potential risks of a new candidate vaccine). Challenge studies with LZ would also provide the opportunity to fully study immunological responses as the sample size is far smaller than that in field efficacy trials; hence one can seek protection correlates that could be used in subsequent vaccine evaluation and selection. Although much is known about immune mechanisms in experimental leishmaniasis, surrogate markers of protective immunity have not been established in humans as of today. It is very difficult and costly to search for such markers in field efficacy trials particularly if children are the target at-risk-population.

In addition, LZ as live challenge in candidate vaccine efficacy trials performed in endemic foci would serve two purposes: a) to evaluate the protective efficacy of the vaccine candidate and b) to protect recipients against naturally occurring CL, usually multiple lesions on the face or other exposed parts of the body. Hence, all participants will be protected, either by the candidate vaccine or by LZ.

Preliminary, safety and immunogenicity trials of LZ:

In preliminary studies as a first step to develop a reproducible challenge system for evaluating various vaccine candidates against leishmaniasis prior to (or possibly instead of) large scale field efficacy trials, frozen live Leishmania major was produced at Razi Institute (5 x 105 promastigotes per inoculation) for use as a live challenge inoculums (19). In a clinical trial to study the safety and immunogenicity of LZ and lesion development resulting from artificial infection, 23 adult male Iranian volunteers were selected and leishmanized (19). Lesion evolution in all volunteers was checked and recorded twice a month and a picture was taken at each follow-up visit until complete healing. Eighty three percent (19/23) of volunteers developed lesions after LZ (17/23 within 60 days of LZ). The largest ulcer size was 17.5 mm. The longest healing period was 285 days (in one volunteer). No serious adverse reaction related to LZ and requiring medical attention was observed or reported. In a second trial, LZ was used in 20 volunteers, including 14 individuals from the first trial (11 had previously developed a lesion and 3 had not). The results demonstrated the similarity between live challenge and natural infection. Indeed, the volunteers who had developed a lesion after the first LZ and the one cured case from natural infection were totally immune and did not develop a new lesion upon live challenge. All volunteers with no history of CL and those who had not developed lesions in the previous trial were not immune and developed a lesion. The course of lesion development was similar to that observed during the first LZ trial. This confirms that LZ can be used effectively and reproducibly as a tool to evaluate the protection induced by a candidate vaccine. In addition, LZ confers immunity to re-infection, should the candidate vaccine fail to do so (19). Subsequent to these studies, a TDR-sponsored, single-blind randomized controlled trial designated LZ3, was performed to assess the safety, immunogenicity and efficacy of four different doses of alum-ALM (10,100, 200 and 320 ug of ALM) plus 1/10th of BCG against CL caused by leishmanization. The target sample size (N = 30 in each arm) was calculated according to 80% power at 0.05 level of confidence, 50% protection against LZ, 60% take rate of LZ in the placebo control group (take rate = lesion development with ulceration) and a 10% loss to follow up. These assumptions were based on the results of two previous leishmanization trials (designated LZ1 and LZ2) in healthy volunteers using the same live parasite (stabilate), which was produced in 1997, standardized and kept frozen in liquid N2 until use. The trial was initiated in 2001 after considerable delay. The time of assessment of efficacy was set at days 135 and 184 (75 and 124 days after live challenge) based on two previous LZ trials using the same stabilate. However, due to the paucity of active lesion development, the protocol was amended to assess the outcome at a later date. This trial suffered from major difficulties. Most importantly, the problems with the live challenge virulence which lead to significantly less-than-expected take rate (about 45% instead of the expected 80-100%), rendered the decided sample size insufficient for vaccine efficacy assessment. However, despite inconclusive efficacy results, this trial clearly demonstrated the safety of different doses of alum-ALM+BCG. To evaluate the efficacy of this candidate vaccine properly, it was decided to repeat the trial.

Risks and Potential Benefits:

As observed in previous trials in Sudan and Iran, risks associated with a single injection of the alum-ALM+BCG are limited to local reactions ranging from induration to ulceration. These lesions are due to the BCG injection used as adjuvant and tend to heal within 30-40 days. Similarly, risks associated with LZ, observed in LZ1, LZ2 and LZ3, are local lesions which heal spontaneously, usually leaving a scar. As stated earlier, LZ as a method of protection is sought after by residents of endemic areas who would otherwise be exposed to a very high chance of natural infection and resulting multiple lesions on face, hands or other exposed parts of the body. In this clinical trial, LZ would lead to protection in individuals who would not be immune as a result of the injection (s) with the candidate vaccine.

Rationale for the trial The clinical trial outlined in this protocol is proposed to evaluate safety, immunogenicity and efficacy of a single and double intradermal injections of 200 ug of Alum-precipitated autoclaved L. major (Alum-ALM) plus BCG vaccine in healthy Iranian volunteers, at high risk of CL due to L. major followed by leishmanization. A comparator group will receive saline in lieu of the candidate vaccine and this group will determine the take rate for the live challenge. Another comparator group will receive BCG in a double-blind manner.

Trial Objectives and Purpose Primary objectives To further evaluate the safety of single- as well as double injections of Alum-ALM (200 ug of Leishmania protein) mixed with 1/10th dose of BCG vaccine within 30 days after booster injection in Iranian volunteers followed by live challenge with L. major for assessment of protection.

To determine the protection induced against live challenge by double injection of Alum-ALM mixed with BCG 30 days after last vaccination.

To determine if a booster injection of Alum-ALM + BCG induces higher immunological responses measured by skin test.

Protection is defined as the absence of ulcerative lesion development (consistent with CL) at Days 180 + 15 after leishmanization at the site of LZ.

Primary endpoints Occurrence of local and/or systemic adverse events (AEs) within 30 days after vaccination assessed by interview, physical examination.

Percentage of volunteers protected against CL (absence of a lesion) compared to controls at day 180 + 15 after LZ.

Dosage regimens Cohort 1. Double injections (30 days apart) of Alum-ALM 200 ug mixed with 1/10 of the normal dose of BCG (n = 50).

Cohort 2. Double injections (30 days apart) of 1/10 of the normal dose of BCG (n = 50).

Cohort 3. Double injections of Comparator (= BCG diluent alone) as control (n = 50) It is expected that all lesions induced by vaccination will be healed before day 60 (day of LZ). All eligible volunteers will receive LZ with the same stabilate on day 60. Volunteers will be monitored for a minimum of 240 days or until the lesions induced by leishmanization are completely healed).

ELIGIBILITY:
Inclusion Criteria:

* Men or women age between 16 to 60 years.
* Generally in good health.
* No known immunological deficiency, including HIV infection (by medical history).
* No fever at the time of vaccination i.e. oral body temperature <37.5°C.
* No history/suspicion/presence of kala-azar or cutaneous leishmaniasis (CL).
* No history of leishmanization.
* No history of vaccination against leishmaniasis.
* No involvement in other drug or vaccine trial(s) during the study period.
* No other known or planned vaccination within 1 month prior to the study and during the study period.
* No current or foreseeable use of immunosuppressors (i.e. corticosteroids) within one month prior to the vaccination and during the period of the study.
* No known allergy to a vaccine component (e.g. BCG, alum hydroxide, etc.).
* Written informed consent provided. If the volunteer is under 18 years old, the legal guardian's signature is required on the informed consent.

Exclusion Criteria:

* Pregnancy.
* Women should not be pregnant and/or lactating and/or planning pregnancy throughout the study period until complete healing of the lesion induced by vaccination and/or leishmanization. A urinary pregnancy test will be performed for all women of child bearing potential at entry and adequate contraception throughout the study should be used if applicable.
* Evidence of prior CL or leishmaniasis (e.g. sign of scar resembling leishmaniasis, confirmed by physical examination).
* Evidence of serious diseases, allergy or allergic conditions leading to medical consultation and treatment especially with steroids or levamisole, recent surgery or hospitalisation, according to the physical examination and medical history interview.
* Presence of any chronic illness/disease including diabetes mellitus, tuberculosis, leprosy, epilepsy and hypertension.
* Abnormal haematology and clinical chemistry (See Sections 8.1.2.1 and 8.1.2.2 for normal ranges of laboratory values).
* Presence of fever at the time of vaccination, i.e. body temperature (by mouth) > 37.5 °C.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2007-01; Primary Completion 2007-05 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Occurrence of local and/or systemic adverse events (AEs) within 30 days after vaccination assessed by interview, physical examination.
Percentage of volunteers protected against CL (absence of a lesion) compared to controls at day 180 + 15 after LZ.

SECONDARY OUTCOMES:
Percentage of volunteers partially protected against CL compared to controls at day 180 + 15 post LZ.
To assess the safety, non expected adverse events after leishmanization, assessed by interview and physical examination (local reactions at the injection site and systemic side effects) until the lesions are completely healed.
In vivo test: Leishmanin skin tests (LST) prior to vaccination (baseline), at Day 23-28 after first injection and at day 52-58 and (before leishmanization) to assess the

CONTACTS AND LOCATIONS:
Overall Officials: Ali Khamesipour, Principal Investigator — Center for Research & Training in Skin Diseases & Leprosy, Tehran University of Medical Sciences; Farrokh Modabber, Study Chair — Center for Research & Training in Skin Diseases & Leprosy, Tehran University of Medical Sciences
Locations (1):
- Center for Research & Training in Skin Diseases & Leprosy, TUMS, Tehran, 14166, Iran

REFERENCES:
- [Background] 1. Lancet 1987; (1): 401-405. 2. New Generation Vaccines, Levine M et al. Eds. Dekker, New York. Chapter 82, 2004. 3. Int J Dermatol. 2002; 41: 73-8. 4. Clinics in Dermat. 14, 5: 489-495, 1996. 5. Clinics in Dermat. 14, 5: 496-502, 1996. 6. The Lancet, 351, 9115:1540-3, 1998. 7. Vaccine, 17, 5: 466-72,1999. 8. Lancet, 356: 1565-69, 2000. 9. Vaccine 2002; 21:174-80 10. J Immunol., 163, 8: 4481-8, 1999. 11. Vaccine, 19: 3485-92, 2001 12. Trans. Roy. Soc. Trop. Med. & Hyg. 97:365-368, 2003 13. J. Exp. Immunol. 2005 (In press). 14. The history of leishmaniasis. Gilles HM, ed. In: Handbook of protozoal infections., Chapman and Hall, 2000. 15. "New developments with human and veterinary vaccine". A Mizrahi, I Hertman, MA Klingberg, A Kohn, eds., Vol. 47, pp. 259-285, Alan R Liss Inc, New York, 1980. 16. Research on Strategies for the Control of Leishmaniasis. Walton, B, Wijeyaretne, PM, Modabber, F. (Eds), International Development Research Center, Ottawa, 336-369, 1988. 17. Bull Soc Fran parasit, 10:183, 1992. 18. Iranian J. Med. Sciences 23, 3&4: 74-80, 1998. 19. Vaccine 23:3642-8, 2005. 20. N Engl J Med. 293,10: 501-2, 1975.